CLINICAL TRIAL: NCT04825483
Title: Effects of a Weight Loss Program in People With Hip Osteoarthritis: a Randomised Controlled Trial
Brief Title: Effects of a Weight Loss Program in People With Hip Osteoarthritis
Acronym: ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20516
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Hip Osteoarthritis; Overweight and Obesity
Keywords: Osteoarthritis; Osteoarthritis, hip; Obesity; Overweight; Weight loss; Arthritis; Joint diseases; Musculoskeletal diseases; Telehealth
MeSH Terms: conditions — Osteoarthritis, Hip; Overweight; Obesity; Osteoarthritis; Weight Loss; Arthritis; Joint Diseases; Musculoskeletal Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A superiority, 2-group, parallel randomised controlled trial
Who Masked: Investigator
Masking Description: Participants will not be informed about the study hypotheses, until the study is completed, at which time they will be provided a lay summary of study findings. However, the components of each treatment arm will be disclosed during recruitment, allowing us to test the interventions in a way whereby potential participants are fully informed about the nature of the components before deciding whether to participate. As the primary and some of the secondary outcomes are participant-reported, participants are also the outcome assessors and are unblinded. Physiotherapists and dietitians will not be blinded to group allocation or study hypothesis. Staff collecting the secondary outcome body composition data will be blinded to group allocation. Research staff administering and entering the participant-reported data will be blinded. Statistical analyses will be performed blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight loss and exercise (Experimental): In addition to the physiotherapist-prescribed exercise program, participants in the weight loss and exercise group will also undergo six consultations with a dietitian. They will undergo a ketogenic very low-calorie diet (VLCD) including meal replacements, with an intensive weight loss phase and weight maintenance phase. The exercise component will be the same as that provided for the exercise only comparator. All dietitian and physiotherapy consultations will be delivered online by video-conference platform.
  Interventions: Other: Weight loss; Other: Exercise
- Exercise only (Active Comparator): Participants will undergo five consultations (30-45 minutes) with a physiotherapist over 6 months for prescription of a home-based strengthening exercise program and physical activity plan (to be conducted independently at home), as well as OA education. All consultations will be conducted remotely via video-conference.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Weight loss — Participants will receive resources to support the weight loss program including a recipe book, activities book and "how-to guide". The diet program comprises two phases: 1) intensive weight loss through a ketogenic Very Low Calorie Diet (VLCD), including meal replacements for two meals/day, and 2) transition from ketogenic VLCD onto a longer-term eating plan for weight maintenance. Meal replacements will be provided free of charge for up to 6 months. Participants will be encouraged to lose at least 10% body weight.
  Arms: Weight loss and exercise
Other: Exercise — Participants will receive resources to facilitate the physiotherapy management plan, including information about the video-conference platform, osteoarthritis information, an exercise plan/log book and a booklet of possible exercises. The physiotherapist consultations include a structured, progressive exercise and physical activity plan. Participants will be given exercise resistance bands and a ankle weight for home exercises.
  Physiotherapists will choose from a list of exercises, aiming to prescribe 5-6 at once. Intensity is determined using a modified Rating of Perceived Exertion (RPE) scale, where it should feel "hard" to "very hard" to perform a full set of each exercises. Participants are encouraged to complete exercises three times per week. Physiotherapists encourage the participant to increase their general and incidental levels of physical/aerobic activity based on their individual needs and goals, as well as their current level of activity.

SUMMARY:
This randomised controlled trial will compare the effects of a weight loss and exercise program to exercise only on clinical outcomes in 100 people with hip osteoarthritis (OA) and overweight or obesity. The primary aim is to find out whether a weight loss and exercise program will improve hip pain more than an exercise program alone at 6 months follow-up

DETAILED DESCRIPTION:
Clinical guidelines recommend exercise as the core treatment for symptoms, but provide conflicting recommendations about weight loss for people with hip OA. Irrefutable health benefits are associated with weight loss for those with overweight or obesity, but it remains uncertain whether weight loss in addition to exercise and regular physical activity is superior to exercise alone for hip OA symptoms.

This study is a randomized controlled trial for which the aim is to determine whether a weight loss and exercise program improves hip pain more than an exercise program alone at 6 months among people with hip OA who have overweight or obesity.

A total of 100 people with hip osteoarthritis and overweight or obesity will be recruited from the community. Participants will be assessed for eligibility, including review of a hip x-ray. They will be enrolled into the study following informed consent and completion of baseline questionnaires and laboratory-based measures. Each participant will be randomly allocated to receive either: a) weight loss plus exercise program or; b) exercise program alone, over 6 months.

The randomisation schedule will be prepared by a biostatistician (permuted block sizes 2 to 6) stratified by site and sex. Participants allocated to the exercise group will be randomly allocated to a physiotherapist. Participants allocated to the exercise plus weight loss group will be randomly allocated to one of the same physiotherapists as the exercise group, and to a dietitian. The schedule will be stored on a password-protected platform at the University of Melbourne and maintained by a researcher not involved in either participant recruitment or administration of outcome measures. Group allocation will be revealed after completion of baseline measures and randomisation.

Dietitians will complete training in best-practice OA management (half day workshop led by investigators), motivational interviewing skills (2-day training course), weight management (the ketogenic very low calorie diet) and trial procedures. Physiotherapists will be trained in trial procedures, best practice OA management, strengthening and physical activity program, behaviour change techniques to promote adherence and resources for use in the program.

Study participants in both groups will attend 5 individual physiotherapy consultations via video-conference over 6 months and will undertake a home-based lower limb muscle strengthening exercise and physical activity program. Those in the weight loss and exercise group will also undertake a ketogenic very low calorie diet (VLCD), which has been demonstrated as a safe and effective means of achieving rapid weight loss in the adult population with overweight/obesity. They will receive meal replacements (maximum 2 per day) for up to 6 months as well as educational resources.

A biostatistician will analyse blinded data. The statistical method will be outlined in a Statistical Analysis Plan.

ELIGIBILITY:
Inclusion Criteria:

* American College of Rheumatology classification criteria with pain in the groin or hip region on most days of the past month and femoral or acetabular osteophytes and joint space narrowing (superior, axial and/ or medial) on x-ray;
* aged 50 years or older;
* report history of hip pain ≥ 3months;
* report an average pain score of at least 4 on an 11-point numeric rating scale (anchored at 0=no pain, 10=worst pain imaginable) over the previous week;
* access to a device with internet connection;
* have a BMI >27 kg/m2;
* willing and able give informed consent and participate fully in the interventions and assessment procedures;
* have ability to weigh themselves (e.g. access to scales);
* pass the Exercise and Sports Science Australia stage 1 adult pre-exercise screening system or obtain general practitioner clearance for participation in the study.

Exclusion Criteria:

* weight >150 kgs (due to the added complexities of additional nutritional requirements for individuals above this weight);
* inability to speak and read English;
* on waiting list for/planning back/lower limb surgery or bariatric surgery in next 12 months;
* previous arthroplasty on affected hip;
* recent hip surgery on affected hip (past 6 months);
* self-reported inflammatory arthritis (e.g. rheumatoid arthritis);
* weight loss of > 2 kg over the previous 3 months;
* already actively trying to lose weight by any of the following mechanisms:

  1. using meal replacements for weight loss
  2. being a member of a commercial weight loss program (e.g. weight watchers)
  3. receiving support from another health care professional for weight loss
  4. using any drugs prescribed to aid in weight loss
  5. using structured meal programs for weight loss such as 'Lite n' Easy'
* unable to undertake ketogenic VLCD without closer medical supervision including self-reported:

  1. diagnosis of Type 1 diabetes
  2. Type 2 diabetes requiring insulin or other medication apart from metformin
  3. warfarin use
  4. stroke or cardiac event in previous 6 months
  5. unstable cardiovascular condition
  6. fluid intake restriction
  7. renal (kidney) problems (unless clearance is obtained from GP, including GP confirmation that estimated glomerular filtration rate >30 mL/min/1.73m2)
* any neurological condition affecting lower limbs;
* pregnancy or planned pregnancy
* vegan dietary requirements due to complexity of delivering a nutritionally complete diet within the ketogenic diet regime.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Severity of hip pain | Change between baseline and 6 months post-randomisation
  Scored on an 11-point Numeric Rating Scale for average hip pain in the last week. Ranges from 0 to 10; where 0=no pain and 10=worst pain possible.

SECONDARY OUTCOMES:
Severity of hip pain | Change between baseline and 12 months post-randomisation
  Scored on an 11-point Numeric Rating Scale for average hip pain in the last week. Ranges from 0 to 10; where 0=no pain and 10=worst pain possible.
Body weight | Change between baseline and 6 months post-randomisation
  Measured on home scales and self-reported in kilograms. The percentage of body weight change (baseline-follow up/baseline x100%) will be calculated .
Body weight | Change between baseline and 12 months post-randomisation
  Measured on home scales and self-reported in kilograms. The percentage of body weight change (baseline-follow up/baseline x100%) will be calculated .
Body Mass Index (BMI) | Change between baseline and 6 months post-randomisation
  Calculated from height and weight, in Kg/m2
Body Mass Index (BMI) | Change between baseline and 12 months post-randomisation
  Calculated from height and weight, in Kg/m2
Total body fat mass | Change between baseline and 6 months post-randomisation
  Measured using dual energy x-ray absorptiometry and reported in grams and % of total body mass
Hip pain | 6 months post-randomisation
  Proportion of participants who meet or exceed the minimal clinical important difference in Numerical Rating Scale for pain (1.8 units). Expressed as percentage relative to number of participants allocated to each group.
Hip pain | 12 months post-randomisation
  Proportion of participants who meet or exceed the minimal clinical important difference in Numerical Rating Scale for pain (1.8 units). Expressed as percentage relative to number of participants allocated to each group.
Hip Osteoarthritis Outcome Scale (HOOS) Pain Subscale | Change between baseline and 6 months post-randomisation
  Scored using 10 questions regarding hip pain in the last week, with Likert response options ranging from no pain to extreme pain. Ranges from 0 to 20 and normalised to 0 - 100 scale. Higher scores indicate less pain.
Hip Osteoarthritis Outcome Scale (HOOS) Pain Subscale | Change between baseline and 12 months post-randomisation
  Scored using 10 questions regarding hip pain in the last week, with Likert response options ranging from no pain to extreme pain. Ranges from 0 to 20 and normalised to 0 - 100 scale. Higher scores indicate less pain.
Hip Osteoarthritis Outcome Scale (HOOS) Activities of daily living subscale | Change between baseline and 6 months post-randomisation
  Scored using 17 questions regarding hip function in the last week, with Likert response options ranging from no dysfunction to extreme dysfunction. Ranges from 0 to 68 and normalised to 0 - 100 scale. Higher scores indicate less dysfunction.
Hip Osteoarthritis Outcome Scale (HOOS) Activities of daily living subscale | Change between baseline and 12 months post-randomisation
  Scored using 17 questions regarding hip function in the last week, with Likert response options ranging from no dysfunction to extreme dysfunction. Ranges from 0 to 68 and normalised to 0 - 100 scale. Higher scores indicate less dysfunction.
Hip Osteoarthritis Outcome Scale (HOOS) Quality of Life Subscale | Change between baseline and 6 months post-randomisation
  Scored using 4 questions regarding quality of life in the last week, with Likert response options ranging from none to extreme. Ranges from 0 to 16 and normalised to 0 - 100 scale. Higher scores indicate better quality of life.
Hip Osteoarthritis Outcome Scale (HOOS) Quality of Life Subscale | Change between baseline and 12 months post-randomisation
  Scored using 4 questions regarding quality of life in the last week, with Likert response options ranging from none to extreme. Ranges from 0 to 16 and normalised to 0 - 100 scale. Higher scores indicate better quality of life.
Quality of life (AQoL-8D) | Change between baseline and 6 months post-randomisation
  Scored from 35 questions regarding health-related quality of life in the last week. Ranges from -0.04 to 1.00; higher scores indicate better quality of life.
Quality of life (AQoL-8D) | Change between baseline and 12 months post-randomisation
  Scored from 35 questions regarding health-related quality of life in the last week. Ranges from -0.04 to 1.00; higher scores indicate better quality of life.
Global rating of change in physical activity | 6 months post-randomisation
  Scored using a 7-point global rating of change Likert scale with response options ranging from "much less" to "much more" when compared to baseline.
Global rating of change in physical activity | 12 months post-randomisation
  Scored using a 7-point global rating of change Likert scale with response options ranging from "much less" to "much more" when compared to baseline.
Global rating of overall change in hip problem | 6 months post-randomisation
  Scored using a 7-point global rating of change Likert scale with response options ranging from "much worse" to "much better" when compared to baseline.
Global rating of overall change in hip problem | 12 months post-randomisation
  Scored using a 7-point global rating of change Likert scale with response options ranging from "much worse" to "much better" when compared to baseline.
Visceral fat mass | Change between baseline and 6 months post-randomisation
  Measured using dual energy x-ray absorptiometry and reported in grams and % of total body mass

CONTACTS AND LOCATIONS:
Overall Officials: Kim Bennell, PhD, Principal Investigator — University of Melbourne
Locations (1):
- University of Melbourne, Carlton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
PD can be shared
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Available upon publication of results
Access Criteria: Upon reasonable request

REFERENCES:
- [Derived] Hall M, Hinman RS, Knox G, Spiers L, McManus F, De Silva AP, Sumithran P, Harris A, Murphy NJ, Cicuttini F, Hunter DJ, Messier SP, Bennell KL. Efficacy of a Very-Low-Calorie Weight Loss Diet Plus Exercise Compared With Exercise Alone on Hip Osteoarthritis Pain : A Randomized Controlled Trial. Ann Intern Med. 2025 Sep;178(9):1227-1237. doi: 10.7326/ANNALS-25-00045. Epub 2025 Aug 5. PMID 40759020
- [Derived] Hall M, Hinman RS, Knox G, Spiers L, Sumithran P, Murphy NJ, McManus F, Lamb KE, Cicuittini F, Hunter DJ, Messier SP, Bennell KL. Effects of adding a diet intervention to exercise on hip osteoarthritis pain: protocol for the ECHO randomized controlled trial. BMC Musculoskelet Disord. 2022 Mar 5;23(1):215. doi: 10.1186/s12891-022-05128-9. PMID 35248012